CLINICAL TRIAL: NCT03288467
Title: Effect of Sodium Hypochlorite Concentration on Success of Non-surgical Root Canal Treatment: A Randomized Controlled Trial.
Brief Title: Effect of Sodium Hypochlorite Concentration on Success of Non-surgical Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neha Verma
Record Dates: First submitted 2017-09-11; First posted 2017-09-20 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2017-09

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Endodontics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment with 5% NaOCl (Active Comparator): Root canal treatment with 5% NaOCl: 5 ml of 5% sodium hypochlorite was used during root canal treatment after each instrument change.After root canal instrumentation, canals irrigated with 5ml of 17% EDTA solution for 1 minute followed by final wash with 5ml of 5% sodium hypochlorite.
  Interventions: Procedure: Root canal treatment with 5% NaOCl
- Root canal treatment with 1% NaOCl (Active Comparator): 5 ml of 1% soium hypochlorite was used during root canal treatment after each instrument change.After root canal instrumentation, canals irrigated with 5ml of 17% EDTA solution for 1 minute followed by final wash with 5ml of 1% sodium hypochlorite.
  Interventions: Procedure: Root canal treatment with 1% NaOCl

INTERVENTIONS:
Procedure: Root canal treatment with 5% NaOCl
  Other Names: Endodontic treatment
  Arms: Root canal treatment with 5% NaOCl
Procedure: Root canal treatment with 1% NaOCl
  Other Names: Endodontic treatment
  Arms: Root canal treatment with 1% NaOCl

SUMMARY:
.There is no general agreement regarding the optimal concentration of sodium hypochlorite to be used in endodontic treatment.Therefore, this study aims to evaluate the effect of sodium hypochlorite concentration on the success of primary root canal treatment. The study population comprised of patients requiring primary root canal treatment following the diagnosis of pulpal necrosis with chronic apical periodontitis in mature mandibular first and second molars.Patients were randomly allocated in either High concentration or Low concentration group.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES

1. To evaluate the success of primary endodontic treatment following use of 5% and 1% NaOCl in non-vital, posterior teeth.
2. To compare the success achieved following use of the two different concentrations of NaOCl.
3. To evaluate postoperative pain following use of 5% and 1% NaOCl.

MATERIALS AND METHODS: Mature mandibular first and second molars with diagnosis of pulp necrosis (as confirmed by negative response to cold and electric pulp testing), and having apical radiolucency were chosen for the study.The consenting subjects were allocated to one of the two study groups based on concentration of NaOCl used: 5% [high concentration (HC)] and 1% [low concentration (LC)].Using an equal proportion randomization allocation ratio, envelopes containing concealed assignment codes were assigned sequentially to eligible patients.It was ensured that neither the patient, nor the primary investigator was aware of the treatment protocol before beginning of the treatment procedure.

CLINICAL PROCEDURE:

2% lidocaine with 1/80000 epinephrine was used to achieve profound local anaesthesia.

After proper isolation with rubber dam, access cavity was made with a high speed handpiece and carbide bur.

Debridement of the pulp chamber was done and all canal orifices were identified Lubricant (RC Prep) was placed at the entrance of the canal and canals negotiated with 10 no. K file.

Working length was established 1mm short of apical foramen by electronic apex loactor (Root ZX) and confirmed radiographically.

Root canal preparation was done by using rotary files according to manufacturer's instructions.

In both groups, 5ml of sodium hypochlorite was used as irrigant after each instrument change. All the irrigation procedures was performed using a 30 gauge needle. 5% and 1% NaOCl was used in HC and LC, respectively.

After root canal instrumentation, canals was irrigated with 5ml of 17% EDTA solution for 1 minute followed by final wash with 5ml of 5% or 1% sodium hypochlorite, depending on the group.

Canals were dried with sterile absorbent paper points and filled with calcium hydroxide paste and the access cavity restored with Cavit.

The patients were recalled after 1 week. At the next appointment, the paste was removed with the use of Hedstroem files and copious irrigation with 5% or 1% sodium hypochlorite followed by 5ml 17% EDTA and a final rinse with 5ml 5% or 1% sodium hypochlorite.

Then, canals were obturated with the Gutta percha by lateral condensation technique and Zinc Oxide- Eugenol based sealer in both the groups.

After obturation, the cavity was restored permanently. Immediate post-operative radiograph was then be taken.

All the patients were prescribed Ibuprofen 400mg with the instructions to take only one tablet every 8 hours in the event of pain, if needed.Patients were asked to record the severity of pain using 10 cm VAS scale with 0 depicting no pain and 10 depicting maximum pain imaginable. Patients were asked to make a mark on the line that represented their level of perceived pain at 6 hr ,12 hr ,1 day,2 days,3 days,4 days,5 days,6 days and 7 days.One week later, patients returned with the completed questionnaires.

Follow up clinical and radiographic examination carried out every 3 months, till 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Patient willingness to participate in the study
* Mature permanent mandibular first and second molars requiring primary root canal treatment
* Diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber
* Radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm)
* Patient's age more than 18 years

Exclusion Criteria

* Positive history of antibiotic use within past one month of the treatment.
* Positive history of analgesic use within the past 3 days.
* Patients who are pregnant, diabetic, immunocompromised, had serious medical illness or required antibiotic premedication
* Patients with pockets ≥4mm or having marginal or furcal bone loss due to periodontitis
* Teeth that are not suitable for rubber dam isolation
* Previously accessed teeth and/or with procedural errors
* Unrestorable tooth, fractured/ perforated roots, inflammatory root resorption

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Radiographic success | Every 3 months till 12 months
  Treatment outcome was judged on the basis of radiographic findings recorded at the follow up visit and comparison of the radiographs obtained at post obturation and the follow-up visit.Change in Periapical Index (PAI) scores observed at 12-months was noted and scoring of each tooth was done according to the PAI scores and score less than 3 were considered as success.
Clinical success | Till 12 months
  Absence of pain and tenderness to palpation/ percussion, absence of sinus or any associated soft tissue swelling, tooth mobility, and no deterioration in periodontal probing depth as compared with baseline measurements comprised the criteria for clinical success.

SECONDARY OUTCOMES:
Pain intensity | Pain intensity recorded at different intervals (preoperatively, after 6 hours, 12 hours, 1day, 2 days, 3 days, 4days, 5 days, 6 days and 7 days).
  Pain intensity before and after treatmemt was recorded by use of 10cm VAS with zero depicting no pain and 10 depicting maximum pain.Patient rate their pain intensity by making a mark somewhere on the line that represents their pain intensity and VAS was scored by measuring the distance from the "no pain" end of line.